CLINICAL TRIAL: NCT01965249
Title: Short Stitch Versus Long Stitch Suture Technique Using Monomax® for Abdominal Wall Closure After Primary Median Laparotomy. A Randomized, Controlled, Double-blinded, Multicenter, International Trial
Brief Title: Effect of Stitch Technique on the Occurrence of Incisional Hernia After Abdominal Wall Closure
Acronym: ESTOIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAG-G-H-1308
Record Dates: First submitted 2013-10-09; First posted 2013-10-18 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Injury of Abdominal Wall
Keywords: Laparotomy; short stitch; long stitch; MonoMax

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Long stitch group (Active Comparator): Long stitch suture technique Stitch interval = 10 mm; Lateral = 10 mm
  Interventions: Device: Long stitch
- Short stitch group (Experimental): Short stitch technique for AWC stitch interval = 5 mm; Lateral 5 - 8 mm
  Interventions: Device: Short Stitch

INTERVENTIONS:
Device: Long stitch — AWC with the long stitch technique using MonoMax USP 1, 150 cm loop, HR48 mm
  Arms: Long stitch group
Device: Short Stitch — Short stitch suture technique using MonoMax USP 2/0, 150 cm, HR26 mm
  Arms: Short stitch group

SUMMARY:
The major long term complication of abdominal wall closure after a median laparotomy is the development of an incisional hernia. Several suture technique and suture material have been used but the incidence of this complication still lies between 9 -20%. Synthetic suture material which have become available over the last decades have the advantage that they are degraded by the body system and fully absorbed within 70-180 days; however they loss 50% of their initial strength already after 14-30 days and may not be the optimal suture material for abdominal wall closure. A new suture material (Monomax®) was developed with an extra-long absorption profile, high elasticity and with a superior initial strength. Therefore, the ESTOIH-Study was designed to investigate the influence of the stitch length on the occurrence of incisional hernia using the extra-long term absorbable, elastic, monofilament suture (Monomax®).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients undergoing an elective, primary median laparotomy with an incision length of ≥ 15 cm
* Expected survival time longer than 1 year
* ASA I-III
* Written informed consent

Exclusion Criteria:

* Emergency surgery
* Patient undergoing surgery due to a pancreas carcinoma
* Patients who will be operated due to an abdominal aortic aneurysm
* Peritonitis
* Coagulopathy
* Current immunosuppressive therapy (more than 40 mg of a corticoid per day or azathioprin)
* Chemotherapy within the last 2 weeks before operation
* Radiotherapy of the abdomen within the last 6 weeks before operation
* Pregnant women (pregnancy test has to be performed)
* Severe neurologic and psychiatric disease
* Lack of compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Incisional hernia rate | 1 year postoperatively
  Incisional hernia rate 1 year postoperatively (assessment by ultrasound).

SECONDARY OUTCOMES:
Frequency of burst abdomen | participants will be followed for the duration of hospital stay, an expected average of 10 days
  Burst abdomen is defined as a clinically evident rupture of the laparotomy wound
Reoperation due to burst abdomen | participants will be followed for the duration of hospital stay, an expected average of 10 days
  Burst abdomen is defined as a clinically evident rupture of the laparotomy wound
Frequency of wound infections | participants will be followed for the duration of hospital stay, an expected average of 10 days and 30 days postop
  Wound infections are classified according to the US centres for disease control and prevention (CDC) as either deep or superficial.
Wound healing complications | until 30 days postoperatively
  Wound healing complications: Seroma, hematoma, necrosis, fistula
Long Term Incisional hernia rate | 3 and 5 years postoperatively
  assessment by ultrasound
Long term Wound infections | 1 year postoperatively
  Wound infections are classified according to the US centres for disease control and prevention (CDC) as either deep or superficial.
Long Term Wound healing complications | until 1 year postoperatively
  Wound healing complications: Seroma, hematoma, necrosis, fistula
Costs | until 5 years postop
  Costs including material cost, cost per operation minute, cost per hospital stay, cost saving per incisional hernia.
Length of postoperative hospital stay | participants will be followed for the duration of hospital stay, an expected average of 10 days
  Number of days the patient has to stay in hospital after the intervention
Course of Health status with EQ-5D Score | preop, 30 days postop, 1 year, 3 years, 5 years postop
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Each answer results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions are combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.

CONTACTS AND LOCATIONS:
Overall Officials: Rene Fortelny, Dr., Principal Investigator — Wilhelminenspital Wien
Locations (9):
- Austria (2):
  - AKH Linz, Linz
  - Wilhelminenspital Wien, Vienna
- Germany (7):
  - Vivantes Klinikum Spandau, Berlin
  - Städtisches Klinikum Braunschweig, Braunschweig
  - Klinikum der Johann-Wolfgang-Goethe Universität, Frankfurt
  - Klinik am Eichert, Allgemeinchirurgische Klinik, Göppingen
  - LMU Großhadern, München
  - Robert Bosch KH Stuttgart, Stuttgart
  - Klinikum Landkreis Tuttlingen, Klinik für Allgemein-, Viszeral, und Gefäßchirurgie, Tuttlingen

REFERENCES:
- [Background] Albertsmeier M, Seiler CM, Fischer L, Baumann P, Husing J, Seidlmayer C, Franck A, Jauch KW, Knaebel HP, Buchler MW. Evaluation of the safety and efficacy of MonoMax(R) suture material for abdominal wall closure after primary midline laparotomy-a controlled prospective multicentre trial: ISSAAC [NCT005725079]. Langenbecks Arch Surg. 2012 Mar;397(3):363-71. doi: 10.1007/s00423-011-0884-6. Epub 2011 Dec 20. PMID 22183105
- [Background] Fischer L, Baumann P, Husing J, Seidlmayer C, Albertsmeier M, Franck A, Luntz S, Seiler CM, Knaebel HP. A historically controlled, single-arm, multi-centre, prospective trial to evaluate the safety and efficacy of MonoMax suture material for abdominal wall closure after primary midline laparotomy. ISSAAC-Trial [NCT005725079]. BMC Surg. 2008 Jul 21;8:12. doi: 10.1186/1471-2482-8-12. PMID 18644124
- [Background] Fortelny RH, Baumann P, Thasler WE, Albertsmeier M, Riedl S, Steurer W, Kewer JL, Shamiyeh A. Effect of suture technique on the occurrence of incisional hernia after elective midline abdominal wall closure: study protocol for a randomized controlled trial. Trials. 2015 Feb 15;16:52. doi: 10.1186/s13063-015-0572-x. PMID 25887884
- [Result] Albertsmeier M, Hofmann A, Baumann P, Riedl S, Reisensohn C, Kewer JL, Hoelderle J, Shamiyeh A, Klugsberger B, Maier TD, Schumacher G, Kockerling F, Pession U, Weniger M, Fortelny RH. Effects of the short-stitch technique for midline abdominal closure: short-term results from the randomised-controlled ESTOIH trial. Hernia. 2022 Feb;26(1):87-95. doi: 10.1007/s10029-021-02410-y. Epub 2021 May 28. PMID 34050419
- [Result] Fortelny RH, Andrade D, Schirren M, Baumann P, Riedl S, Reisensohn C, Kewer JL, Hoelderle J, Shamiyeh A, Klugsberger B, Maier TD, Schumacher G, Kockerling F, Pession U, Hofmann A, Albertsmeier M. Effects of the short stitch technique for midline abdominal closure on incisional hernia (ESTOIH): randomized clinical trial. Br J Surg. 2022 Aug 16;109(9):839-845. doi: 10.1093/bjs/znac194. PMID 35707932
- [Result] Fortelny RH, Hofmann A, Baumann P, Riedl S, Kewer JL, Hoelderle J, Shamiyeh A, Klugsberger B, Maier TD, Schumacher G, Kockerling F, Pession U, Schirren M, Albertsmeier M. Three-year follow-up analysis of the short-stitch versus long-stitch technique for elective midline abdominal closure randomized-controlled (ESTOIH) trial. Hernia. 2024 Aug;28(4):1283-1291. doi: 10.1007/s10029-024-03025-9. Epub 2024 Mar 27. PMID 38536592
- [Result] Fortelny RH, Baumann P, Hofmann A, Riedl S, Kewer JL, Hoelderle J, Shamiyeh A, Klugsberger B, Maier TD, Schumacher G, Kockerling F, Woste G, Pession U, Albertsmeier M. 5-year clinical outcome of the ESTOIH trial comparing the short-bite versus large-bite technique for elective midline abdominal closure. Hernia. 2025 Aug 29;29(1):263. doi: 10.1007/s10029-025-03459-9. PMID 40879826